CLINICAL TRIAL: NCT04069871
Title: Effect of Transcutaneous Electrical Nerve Stimulation on Tissue Perfusion for the Critically Ill Patient
Brief Title: Transcutaneous Electrical Nerve Stimulation for Tissues Perfusion
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mostafa Samy Abbas, associate professor of anesthesia, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: TENS
Record Dates: First submitted 2019-08-23; First posted 2019-08-28 (Actual); Last update posted 2020-12-16 (Actual); Status verified 2020-12

CONDITIONS: Renal Function Disorder; Critical Illness; Critical Illness Myopathy
MeSH Terms: conditions — Critical Illness

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TENS (Active Comparator)
  Interventions: Device: trans-cutaneous electrical nerve stimulation.
- Control (Sham Comparator)
  Interventions: Device: Sham TENS

INTERVENTIONS:
Device: trans-cutaneous electrical nerve stimulation. — • Patients assigned to the EMS group received daily EMS sessions of both lower extremities starting from the second day for 5days.
  Arms: TENS
Device: Sham TENS — Patients in the control group will receive sham TENS.
  Arms: Control

SUMMARY:
The aim of this study is to determine the effect of transcutaneous electrical nerve stimulation in mechanically ventilated patients on the lower limb and renal tissue perfusion.

ELIGIBILITY:
Inclusion Criteria:

* Recently intubated patient.
* Adult and both gender.
* Hemodynamic stability

Exclusion Criteria:

* Vascular diseases
* Diabetic patients
* Patients who receive vasoactive drugs
* Patients with varicose vein
* Systemic scoliosis

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2019-10-15 (Actual); Primary Completion 2020-10-06 (Actual); Study Completion 2020-10-06 (Actual)

PRIMARY OUTCOMES:
tissue perfusion of the lower limb. | 5 ICU days
  capillary refill time
Renal perfusion | 5 ICU days
  quantitative assessment of neutrophil gelatinase-associated lipocalin

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut University hospital, Asyut, Asyut Governorate, Egypt